CLINICAL TRIAL: NCT04871880
Title: Lifestyle Modification for the Treatment of Metabolic Associated Fatty Liver Disease Based on Transtheoretical Model: a Single-center, Randomized, Controlled Study
Brief Title: Lifestyle Modification for MAFLD Based on TTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2019-254
Record Dates: First submitted 2021-04-20; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Associated Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietitian led life style modification intervention. (Experimental): Lifestyle changes supervised by dietitians
  Interventions: Behavioral: Dietitian led life style modification intervention
- Conventional care (control) (Experimental): Receive routine care
  Interventions: Behavioral: Conventional care (control)

INTERVENTIONS:
Behavioral: Dietitian led life style modification intervention — All participants received recommendations for a low-fat hypocaloric diet that was 750 kcal/day less than their daily energy need which supervised by dietitians. Additionally, patients were encouraged to walk 200 minutes per weeks and a short self-report questionnaire for the measurement of habitual physical activity was implemented at baseline, 4, 16, 32 and 48 weeks.
  Arms: Dietitian led life style modification intervention.
Behavioral: Conventional care (control) — Receive routine care
  Arms: Conventional care (control)

SUMMARY:
Lifestyle changes aiming at weight loss remain the cornerstone of MAFLD treatment.Evaluating the motivational stage of patients' change and providing targeted lifestyle guidance may significantly improve the efficiency of weight loss. The investigators hypothesize that gut microbiota may affect motivation to lose weight, and the changes in gut microbiota due to weight loss may positively feedback the behavior of motivation, forming a virtuous circle. Thus, this study aims at ①evaluating the relationships between motivational stage of weight loss and the gut microbiota (Gut-brain axis); ②investigating the effects of lifestyle interventions on the gut microbiota in MAFLD patients.

DETAILED DESCRIPTION:
Fatty liver associated with metabolic dysfunction is common, affects a quarter of the population, and has no approved drug therapy. In 2020, two position articles have proposed not only the change of the terminology from NAFLD to metabolic associated fatty liver disease (MAFLD), but also an update and revision of the definition of fatty liver disease. According to these papers, indeed, the diagnosis of MAFLD can be made with the presence of hepatic steatosis (detected by serum biomarker scores, imaging methods or histology) and at least one of the fol- lowing metabolic criteria: (a) overweight/obesity, (b) T2DM and (c) metabolic dysregulation (that means at least two factors among increased waist circumference, hypertension, hypertriglyceridemia, low serum HDL-cholesterol levels, impaired fasting glucose, homeostatic model assessment of insulin resistance [HOMA-IR] > 2.5 or high sensitivity C-reactive protein > 2 mg/L). Here，the investigators focus on the obese NAFLD, which considered as a sub-phenotype in MAFLD.

Lifestyle changes aiming at weight loss remain the cornerstone of MAFLD treatment. However, it is not easy to make patients change their unhealthy lifestyle. Behavior therapy may only be successful in motivated patients, and motivation to dieting and exercising may be different according to age and sex. Personal motivation for change plays a pivotal role in behavior changes. The transtheoretical model (TTM) is an empirically validated model of individual behavioral change, which involves progress through a series of stages to make a particular behavioral change. TTM-based interventions have been applied to facilitate health behavioral changes, such as physical exercise, smoking cessation, and weight management, studies of which continue to demonstrate positive effects. Evaluating the motivational stage of patients' change and providing targeted lifestyle guidance may significantly improve the efficiency of weight loss. The investigators hypothesize that gut microbiota may affect motivation to lose weight, and the changes in gut microbiota due to weight loss may positively feedback the behavior of motivation, forming a virtuous circle.

Thus, a total of seventy obese patients with NAFLD will be recruited in this study, divided into lifestyle modification program group(n=35) and usual care group(n=35). All subjects will undergo dietary assessment based on Food Frequency Questionnaire ( FFQ) and motivational stages evaluation based on TTM. Stool samples will be collected at each visit. Demographic data will be recorded, consisted of age, weight, height, waist circumference, BMI, and so on. MRI-PDFF will be performed to evaluate liver steatosis. Meanwhile, vibration-controlled transient elastography will be carried out, which include liver stiffness (LSM) and controlled attenuation parameter (CAP) measurements. Biochemistry tests will be conducted as supplementary for assessment of NAFLD and cardiovascular risks, comprising liver function test, lipid, fasting glucose, etc.

The investigators aim at ①evaluating the relationships between motivational stage of weight loss and the gut microbiota (Gut-brain axis); ②investigating the effects of lifestyle interventions on the gut microbiota in MAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

1. With age range of 18-65 years.
2. BMI ≥ 28kg/m2
3. Fatty infiltration of the liver was confirmed on imaging studies (ultrasound, transient elastography, computed tomography, or magnetic resonance imaging) or liver biopsy.
4. With valid motivational stage assessment based on TTM.
5. Written consent form obtained.

Exclusion Criteria:

1. History of other chronic liver disease (Viral hepatitis B or C, autoimmune hepatitis, cholestatic and Inherited metabolic liver diseases) and hemochromatosis.
2. Self-reported HIV-positive status, active tuberculosis, active malaria, or inflammatory bowel disease.
3. Excessive alcohol consumption (>30g/d for men and >20g/d for women).
4. Patient has known cirrhosis (compensated/decompensated) either based on clinical criteria or liver histology or Imaging techniques.
5. Subjects using thyroid hormones, oestrogens, amiodarone, steroids, tamoxifen and other medicine known to affect liver fat accumulation.
6. Subjects using thiazolidinedione hypoglycemic drugs, vitamin E and other medicine have potential benefits for NASH within six months.
7. Subjects with organ failure.
8. Subjects with hepatocellular carcinoma or other active malignancy.
9. Solid organ transplant recipients.
10. Antibiotic treatment within the previous 3 months.
11. Suffering from any acute or chronic cardiovascular, GI or immunological condition.
12. Gastric or duodenal ulcer in the past six months.
13. Currently pregnant or nursing.
14. Concomitant diseases with reduced life expectancy.
15. Combined mental illness.
16. Contraindication to MRI scanning.
17. Exclusions may also be made at the discretion of the attending physician or the eligibility committee.
18. Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Hepatic fat | 12 months
  Change of liver proton density fat fraction (PDFF) in MAFLD assessed by magnetic resonance imaging (MRI)
Obesity | 1, 4, 8, 12, 24 months
  Changes in body weight
Gut microbiota | 1, 4, 8, 12, 24 months
  Changes in bacterial component of the gut microbiome

SECONDARY OUTCOMES:
Blood pressure | 1, 4, 8, 12, 24 months
  Changes in blood pressure
Central obesity | 1, 4, 8, 12, 24 months
  Changes in waist circumference
Insulin resistance | 1, 4, 8, 12, 24 months
  Changes in insulin resistance eveluated by HOMA-IR
FPG | 1, 4, 8, 12, 24 months
  Changes in fast plasma glucose
HbA1c | 1, 4, 8, 12, 24 months
  Changes in HbA1c
Plasma triglycerides | 1, 4, 8, 12, 24 months
  Changes in plasma triglycerides
Plasma HDL-cholesterol | 1, 4, 8, 12, 24 months
  Changes in plasma HDL-cholesterol
Plasma high-sensitivity C-reactive protein level | 1, 4, 8, 12, 24 months
  Changes in plasma high-sensitivity C-reactive protein level
Gut microbiota diversity | 1, 4, 8, 12, 24 months
  Changes in diversity of gut microbiome(α-diversity and β-diversity)

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided